CLINICAL TRIAL: NCT02363517
Title: The Treatment And Prevention (TAP) Study: Treating People Who Inject Drugs (PWID) in Community-based Settings Using a Social Network Approach
Brief Title: The TAP Study: Treating People Who Inject Drugs in Community-Based Settings Using a Social Network Approach
Acronym: TAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: St Vincent's Hospital Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MacfarlaneBIMRPH
Record Dates: First submitted 2014-12-21; First posted 2015-02-16 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis C; Drug Abuse, Intravenous
Keywords: Hepatitis; Viral; Non-A; Non-B; Parenterally-Transmitted
MeSH Terms: conditions — Hepatitis C; Substance Abuse, Intravenous; Hepatitis | interventions — Sofosbuvir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (No Intervention): Primary (n=40) and secondary (n=100) participants will receive supportive care only (includes a clinical review, questionnaire and blood sample collected at baseline and weeks 12, 24, 36, 48, 60, 72 and 84).
  Participants with HCV not allocated to treatment arms will receive deferred treatment at the end of the follow-up period.
- Group B (Active Comparator): Primary participants (n=40) will be treated with 'Sofosbuvir/ledispasvir fixed dose combination (SOF + LDP) for 12 weeks. Secondary participants (n=100) will receive supportive care only.
  Participants with HCV not allocated to treatment arms will receive deferred treatment at the end of the follow-up period.
  Interventions: Drug: Sofosbuvir/ledispasvir fixed dose combination (SOF + LDP)
- Group C (Active Comparator): Primary (n=40) and secondary participants with chronic HCV infection (approx. n=50%*100) will be treated with 'Sofosbuvir/ledispasvir fixed dose combination (SOF + LDP) for 12 weeks. Participants in Group C who have evidence of HCV re-infection will be offered re-treatment with SOF + LDP for 12 weeks.
  Interventions: Drug: Sofosbuvir/ledispasvir fixed dose combination (SOF + LDP)

INTERVENTIONS:
Drug: Sofosbuvir/ledispasvir fixed dose combination (SOF + LDP) — SOF + LDV tablets contain 400mg of SOF and 90mg of LDV.
  Other Names: Standard of care
  Arms: Group B; Group C

SUMMARY:
This study will investigate the feasibility of treating people who inject drugs (PWID) with hepatitis C virus (HCV) in community-based settings with a 12-week course of oral therapy combination of sofosbuvir plus ledipasvir. It will also measure the effectiveness of using a social network-based approach to reduce HCV incidence among PWID.

DETAILED DESCRIPTION:
This study will investigate the feasibility of treating people who inject drugs (PWID) with hepatitis C virus (HCV) in community-based settings with a 12-week course of oral therapy combination of sofosbuvir plus ledipasvir (SOF + LDP). It will also measure the effectiveness of using a social network-based approach ("bring your friends") to reduce HCV incidence among PWID. Participants will initially be sourced from the Burnet Institute's existing SuperMIX cohort (N= 757). This cohort comprises PWID followed for between two and six years (median=1057 days), of whom 299 have chronic HCV infection. The HCV genotype distribution in the SuperMIX cohort is: HCV-1 (55%); HCV-3 (40%) and HCV-6 (<5%).

Participants will be randomly allocated to three groups:

Group 1: Primary (n=40) and secondary (n=100) participants will receive supportive care only.

Group 2: Primary participants (n=40) will be treated with SOF + LDP for 12 weeks. Secondary participants (n=100) will receive supportive care only.

Group 3: Primary (n=40) and secondary participants with chronic HCV infection (n=50%*100) will be treated with SOF + LDP for 12 weeks. Participants in Group C who have evidence of HCV re-infection will be offered re-treatment with SOF + LDP for 12 weeks.

Treatment participants will have a clinical review, questionnaire and blood sample collected at baseline, weeks 4, 8 and 12 (end-of-treatment), and at weeks 12 (SVR12), 24 (SVR24), 36, 48, 60 and 72 post-treatment. Non-treatment participants will have a clinical review, questionnaire and blood sample collected at baseline and weeks 12, 24, 36, 48, 60, 72 and 84.

ELIGIBILITY:
SECONDARY PARTICIPANTS INCLUSION AND EXCLUSION CRITERIA

Study INCLUSION criteria for primary participants are as follows:

* Current PWID (i.e., injected any drug at least once during the previous six months);
* Evidence of chronic HCV infection (detectable plasma HCV RNA viral load above 1000 IU/ml on two occasions ≥ 6 months apart)
* Willing and able to provide written informed consent.

Subjects must have the following laboratory parameters at screening:

* ALT <10 times the upper limit of normal (ULN)
* AST <10 times ULN
* Haemoglobin ≥12g/dL for males, ≥11g/dL for female subjects
* INR ≤1.5 times ULN unless is stable on an anticoagulant regimen affecting INR
* Albumin ≥3g/dL
* Direct bilirubin ≤1.5 times ULN
* Creatinine clearance (CLcr) ≥60mL/min, as calculated by the Cockcroft-Gault Equation.

EXCLUSION criteria for all primary participants are as follows:

* Testing positive for HIV
* History of, or current, decompensated liver disease
* Testing positive for HBsAg
* HCC
* Women who are pregnant or breastfeeding, or men with female partners who are pregnant at screening or baseline, or who were pregnant in the six months prior to screening
* Already enrolled in the TAP Study as a secondary participant (see below)
* Evidence of any condition, therapy, laboratory abnormality or other circumstance (current or prior) that may confound the study's results, or interfere with participation for the full duration of the study, such that it is not in the best interest of the participant;
* Use of concomitant medications.

Additional EXCLUSION criteria for primary participants with HCV genotypes 2-6:

* Increased baseline risk for anaemia (e.g., a history of thalassemia, spherocytosis, history of GI bleeding), or for whom anaemia would be medically problematic;
* Documented or presumed coronary artery disease or cerebrovascular disease if, in the judgment of the investigator, an acute decrease in haemoglobin by up to 4g/dL (as may be seen with ribavirin therapy) would not be well-tolerated.

SECONDARY PARTICIPANTS INCLUSION AND EXCLUSION CRITERIA

The INCLUSION criteria for secondary participants are as follows:

* Is nominated by a primary participant as a current injecting partner (i.e., has engaged in IDU with a primary participant in the previous six months)
* Willing and able to provide written informed consent.

There are no exclusion criteria for secondary participants who are not receiving HCV therapy in this protocol:

EXCLUSION criteria for treated secondary participants (i.e., those in Group C who are HCV positive) are as follows:

* History of, or current, decompensated liver disease
* Women who are pregnant or breastfeeding, or men with female partners who are pregnant at screening or baseline, or who were pregnant in the six months prior to screening
* Testing positive for HIV
* Testing positive for HBsAg
* HCC
* Evidence of any condition, therapy, laboratory abnormality or other circumstance (current or prior) that may confound the study's results, or interfere with participation for the full duration of the study, such that it is not in the best interest of the participant
* Use of concomitant medications.

Additional EXCLUSION criteria for secondary participants with HCV genotypes 2-6:

* Increased baseline risk for anaemia (e.g. a history of thalassemia, spherocytosis, history of GI bleeding) or for whom anaemia would be medically problematic
* Documented or presumed coronary artery disease or cerebrovascular disease if, in the judgment of the investigator, an acute decrease in haemoglobin by up to 4g/dL (as may be seen with ribavirin therapy) would not be well-tolerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of treating PWID with HCV using 12 weeks of oral therapy via a community-based, nurse-led treatment model, as measured by SVR rates | Change in sustained viral response rates at weeks 12 and 24 post-treatment. Participant retention rate at weeks 4, 8 and 12 (end of treatment).
The effectiveness of treating PWID on rates of HCV primary infection and reinfection among their social networks, as measured by HCV incidence rates among primary and secondary participants | Changes in rates of HCV primary infection and reinfection at weeks 12, 24, 36, 48, 60, 72 and 84
  Hypothesis: Offering HCV treatment to PWID will lead to a lower incidence of transmission of HCV from primary participants to their injecting partners, compared to not treating any PWID.
The effectiveness of treating PWID using a "bring your friends" strategy on rates of HCV primary infection and reinfection, as measured by HCV incidence rates among participants | Changes in rates of HCV primary infection and reinfection at weeks 12, 24, 36, 48, 60, 72 and 84
The feasibility of treating PWID with HCV using 12 weeks of oral therapy via a community-based, nurse-led treatment model, as measured by SVR rates and participant retention | Change in participant retention rates at weeks 4, 8 and 12 (end of treatment)

SECONDARY OUTCOMES:
Changes in levels of injecting risk behaviours among participants following HCV treatment, as measured by self-reported frequency of risky injecting behaviours among participants | Weeks 12, 24, 36, 48, 60, 72 and 84
Changes to Quality of Life (QoL) among treated participants versus non-treated participants, as measured by self-reported responses to validated QoL scales | Weeks 12, 24, 36, 48, 60, 72 and 84
The prevalence of HCV resistance associated variants among treated participants who do not achieve SVR12 | At 12 weeks post-treatment (SVR12) and weeks 24 (SVR24), 36, 48, 60 and 72 post-treatment
Changes in the level of transient liver elastography readings (measured using Fibroscan®) among treated participants versus non-treated participants | Up to 84 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof Margaret Hellard, Principal Investigator — Burnet Institute; Prof Alexander Thompson, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- Burnet Institute, Melbourne, Victoria, Australia